CLINICAL TRIAL: NCT03516136
Title: A Retrospective Study for Collecting Data on the Safety and Performance of the EndoFast Reliant SCP in Vaginal Wall Reinforcement
Brief Title: Safety and Performance of the EndoFast Reliant SCP in Vaginal Wall Reinforcement
Status: Completed | Type: Observational
Sponsor: Allium, Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: CL-SCP-60-04-R
Record Dates: First submitted 2018-04-03; First posted 2018-05-04 (Actual); Last update posted 2018-05-17 (Actual); Status verified 2018-04

CONDITIONS: Pelvic Organ Prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Device: No

INTERVENTIONS:
Device: EndoFast Reliant SCP — POP repair procedure with the EndoFast Reliant SCP system

SUMMARY:
A Single arm, single site, retrospective cohort Post Marketing Clinical Follow up Study Evaluating the Safety and Performance of the EndoFast Reliant SCP for apical support.

ELIGIBILITY:
Inclusion Criteria:

1. Female subjects >18 years old that underwent Pelvic Organ Prolapse repair utilizing the EndoFast Reliant SCP

Exclusion Criteria:

1. Patients without follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All Female subjects >18 years old that underwent Pelvic Organ Prolapse repair utilizing the EndoFast Reliant SCP
Sampling Method: Non-Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-12-31 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Safety- procedure and device related complication rate | Up to 4 years
  Percentage of device and procedure related complications.

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol (2017-03-13): https://cdn.clinicaltrials.gov/large-docs/36/NCT03516136/Prot_001.pdf